CLINICAL TRIAL: NCT06495216
Title: Exploratory Safety and Effectiveness Evaluation of Pulsed Field Ablation by a Balloon Catheter With the TRUPULSE Generator for Treatment of Paroxysmal Atrial Fibrillation (PAF)
Brief Title: Exploratory Safety and Effectiveness Evaluation of Pulsed Field Ablation (PFA) by Balloon Catheter With TRUPULSE Generator for Treatment of Paroxysmal Atrial Fibrillation (PAF)
Acronym: ZephIRE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision; no sites were activated nor were any patients enrolled
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWI202304
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulsed Field Ablation by a Balloon Catheter with the TRUPULSE Generator (Experimental): Participants with paroxysmal atrial fibrillation (PAF) will undergo pulmonary vein (PV) ablation procedure with investigational system (pulsed field ablation balloon catheter used in combination with the TRUPULSE generator) until pulmonary vein isolation (PVI) is achieved and confirmed via entrance block. If PVI cannot be achieved with the investigational system, a commercially approved Biosense Webster (recommended) catheter and compatible commercially available generator can be used to complete the procedure.
  Interventions: Device: Pulsed Field Ablation by a Balloon Catheter with the TRUPULSE Generator

INTERVENTIONS:
Device: Pulsed Field Ablation by a Balloon Catheter with the TRUPULSE Generator — Pulsed field ablation balloon catheter and TRUPULSE generator will be used for PV ablation.

SUMMARY:
The purpose of this study is to explore preliminary safety and acute effectiveness of pulsed field ablation by the ablation system (pulsed field ablation balloon catheter and TRUPULSE generator) when used for isolation of the atrial pulmonary veins (PVs) in treatment of participants with paroxysmal atrial fibrillation (PAF), an irregular heart rate that causes abnormal blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with symptomatic Paroxysmal Atrial Fibrillation (PAF) defined as AF that terminates spontaneously or with intervention within 7 days of onset. This PAF is considered to be symptomatic if symptoms related to AF are experienced by the participant
* Selected for AF ablation procedure by pulmonary vein isolation (PVI)
* Willing and capable of providing consent
* Able and willing to comply with all pre-, post-, and follow-up testing and requirements

Exclusion Criteria:

* Previously known AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause (example, documented obstructive sleep apnea, acute alcohol toxicity, morbid obesity [body mass index more than {>} 40 kilogram per square meter {kg/m^2}], renal insufficiency [with an estimated creatinine clearance less than {<}30 milliliter {mL}/minute {min}/1.73 meter {m}^2])
* Previous left atrium (LA) ablation or surgery
* Participants known to require ablation outside the pulmonary vein (PV) region (example, atrioventricular reentrant tachycardia, atrioventricular nodal re-entry tachycardia, atrial tachycardia, ventricular tachycardia and Wolff-Parkinson-White)
* Previously diagnosed with persistent AF (>7 days in duration)
* Severe dilatation of the LA (left anterior descending artery [LAD] >50 millimetre [mm] antero-posterior diameter or left atrium volume index [LAVi] >48 [mL/m^2] in case of transthoracic echocardiography [TTE])

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-17 (Estimated); Primary Completion 2025-03-26 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Primary Adverse Events (PAEs) | Up to 3 months post-procedure
  Percentage of participants with PAEs will be reported. PAE's will include the following adverse events: atrio-esophageal fistula, phrenic nerve paralysis, cardiac tamponade/perforation, severe pulmonary vein stenosis (PVS), device or procedure related death, stroke/cerebrovascular accident (CVA), major vascular access complication/bleeding, thromboembolism, myocardial infarction, transient ischemic attack (TIA), pericarditis, heart block, pulmonary edema (respiratory insufficiency), and vagal nerve injury/gastroparesis.
Percentage of Participants with Acute Effectiveness | Up to 3 months post-procedure
  Percentage of participants with acute effectiveness will be reported. Acute effectiveness is an electrical isolation of clinically relevant targeted pulmonary veins (PVs) which is evidenced by confirmation of entrance block, after adenosine/isoproterenol challenge, at the end of the index ablation procedure.

SECONDARY OUTCOMES:
Percentage of Participants with Freedom from Documented (Symptomatic and Asymptomatic) Atrial Arrhythmia (Atrial Fibrillation [AF], Atrial Tachycardia [AT] or Atrial Flutter [AFL] of Unknown Origin) Episodes During the Effectiveness Evaluation Period | Within Day 91 to Day 365
  Percentage of participants with freedom from documented (symptomatic and asymptomatic) atrial arrhythmia (AF, AT or AFL of unknown origin) episodes based on electrocardiographic data (more than equal to [>=]30 seconds on arrhythmia monitoring device) during the effectiveness evaluation period (Day 91 to Day 365) on or off antiarrhythmic therapy will be reported. Acute procedural failure (that is, failure to achieve entrance block with the study device in any of the clinically relevant targeted PVs) will also be deemed a 12-month effectiveness failure.
Percentage of PVs that are Targeted in the Index Ablation Procedure with Sustained Isolation at Day 75 | Day 75
  Percentage of PVs that are targeted in the index ablation procedure with sustained isolation, which is evidenced by electrical confirmation (through pacing for entrance block) of isolation at Day 75 post index ablation procedure will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Biosense Webster, Inc. Clinical Trial, Study Director — Biosense Webster, Inc.

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu